CLINICAL TRIAL: NCT06793111
Title: Visceral Leishmaniasis in Emilia-Romagna
Brief Title: Visceral Leishmaniasis in Emilia-Romagna (Leishmania-2019)
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: AUSL Romagna Rimini (Other); Ospedale Bufalini di Cesena, Italy (Unknown); Morgagni Pierantoni Hospital (Other); Ospedale "Santa Maria delle Croci" di Ravenna - AUSL Romagna (Unknown)
Responsible Party: Sponsor
Other Study IDs: Leishmania-2019
Record Dates: First submitted 2024-12-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Leishmaniasis, Visceral
Keywords: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to reports in the literature, from 2012 to date, there has been an increase in the number of diagnosed cases of autochthonous visceral Leishmania in the Province of Bologna.

In this context, it was decided to carry out a retrospective prospective observational study, which is essential to describe the epidemiology of LV in order to outline the scientific and rational bases necessary for the drafting of guidelines to standardise the diagnostic and therapeutic approach to this disease, in order to reduce the diagnostic delay and improve therapeutic results.

therapeutic outcome. In addition, epidemiological data will make it possible to identify possible new strategies to control the disease, which are essential for reducing its transmission.

DETAILED DESCRIPTION:
The term leishmaniasis refers to a heterogeneous group of anthropo-zoonoses caused by protozoa obligate intracellular protozoa, parasites of humans and various wild and domestic animals, belonging to the genus Leishmania. Despite being the cause of recurrent epidemic outbreaks with high rates of morbidity and mortality rates in certain geographical areas, the World Health Organisation (WHO) includes them among the Neglected Tropical Diseases. About 350 million people live in areas at risk for leishmaniasis with an estimated global prevalence of 12 million. The annual global incidence is estimated to be between 0.2 and 0.4 million cases for Visceral Leishmaniasis (LV) and between 0.7 and 1.2 million cases for Cutaneous Leishmaniasis Cutaneous. Leishmaniases are endemic infections in tropical, subtropical and temperate zones of all continents except Australia and Antarctica. More than 90% of LV cases are diagnosed in six countries: Bangladesh, Brazil, Ethiopia, India, South Sudan and Sudan, while the majority of LC cases are diagnosed in Afghanistan, Algeria, Brazil, Colombia, Iran, Pakistan, Peru, Saudi Arabia and Syria.

Leishmaniasis is also endemic in the Mediterranean Basin, including Italy, and in this area about 5% of global cases are found there, with a clear prevalence of visceral forms.

The incubation period varies from 4 to 10 months, but cases have been described in which incubation lasted for several years.

The onset is mostly gradual and insidious and the most characteristic clinical manifestations are asthenia fever (often initially framed as FUO), night sweats, anorexia and weight loss, splenomegaly, hepatomegaly and lymphadenomegaly. From a laboratory point of view, characteristic are anaemia, leucopenia and thrombocytopenia, more or less associated with each other, up to full-blown pancytopenia.

Dysprotidemia with hypergammaglobulinemia and hypoalbuminemia is typical. If not adequately treated, visceral leishmaniasis evolves towards a condition of cachexia and profound general decay and may prove fatal. A rare and serious complication of LV is the haemophagocytic syndrome. According to the 2010 WHO Leishmaniasis Control Report, a confirmed case of LV is defined as the association between typical clinical signs and symptoms (fever, splenomegaly, weight loss, etc.) and positivity of a parasitological examination (microscopy, RT-PCR or culture) in the presence or absence of positivity of serological investigations.

The methods available for the diagnosis of LV include:

* Serological tests: detection of Leishmania-specific IgG (or total Ig) in plasma or serum. enzyme immunoassay (EIA), indirect immunofluorescence assay (IFAT), immunochromatographic test (ICT) based on the immunochromatographic test (ICT) based on rK39 antigen, Western blot (WB). Disadvantages: these tests remain positive over time (it is not always possible to distinguish relapses); they may be positive in individuals with asymptomatic infection; they may be falsely negative in immunodepressed individuals (20-60% of cases).
* Molecular biology tests: detection of Leishmania DNA by RT-PCR on peripheral blood bone marrow blood or any other material. Molecular tests are now considered the most sensitive methods sensitive for the diagnosis of LV and the accuracy in identifying Leishmania DNA is high for bone marrow aspirate and peripheral blood samples. RT-PCR should be performed in case the presence of suspicious symptoms and serological test positivity. However, in the presence of strong suspicion clinical suspicion or in immunocompromised patients, RT-PCR should also be performed in case of a negative serology test.

Quantitative RT-PCR on peripheral blood may be useful in patients immunocompromised patients for monitoring parasitukaemia during therapy.

Direct microscopic examination on bone marrow blood smear: sensitivity is variable (25-85%) and lower than the sensitivity of molecular methods.

- Culture examination: culture isolation from bone marrow blood takes a long time (at least 4 weeks). Culture allows the isolation of the strain of Leishmania responsible for the disease and can also be can also be performed from biopsy tissue.

According to reports in the literature, from 2012 to date, there has been an increase in the number of diagnosed cases of autochthonous visceral Leishmania in the Province of Bologna.

In this context, it was decided to carry out a retrospective prospective observational study, which is essential to describe the epidemiology of LV in order to outline the scientific and rational bases necessary for the drafting of guidelines to standardise the diagnostic and therapeutic approach to this disease, in order to reduce the diagnostic delay and improve therapeutic results.

therapeutic outcome. In addition, epidemiological data will make it possible to identify possible new strategies to control the disease, which are essential for reducing its transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with microbiologically established diagnosis of LV.
* Obtaining Informed Consent.

Exclusion Criteria:

* not having obtained Informed Consent

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a diagnosis of established Visceral Leishmaniasis but also patients with a diagnosis of prior Visceral Leishmaniasis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of Visceral Leishmaniasis (VL) cases in Emilia-Romagna | March 2020 - February 2025
  In-depth description of the epidemiology of autochthonous visceral Leishmaniasis in the Emilia-Romagna region, focusing on the increase in diagnosed cases since 2012. The study will provide critical data for identifying trends in incidence, affected populations, and geographical hotspots, essential for guiding public health interventions.
  Measure: Number of diagnosed cases per year across participating centers. Unit of measure: Number of cases (n). Collection method: Review of medical records and epidemiological registries.
Socio-demographic and clinical characteristics of patients diagnosed with VL | March 2020 - February 2025
  Detailed analysis of the clinical features and presentations of diagnosed LV cases, including common symptoms such as fever, weight loss, splenomegaly, and laboratory findings like anemia and pancytopenia. This analysis will help establish a clearer clinical profile for early diagnosis and treatment strategies.
  Measure: Age, gender, comorbidities, geographic area of residence, known exposure mode.
  Unit of measure: Mean ± standard deviation (continuous variables), percentages (categorical variables).
  Collection method: clinical data collection.

SECONDARY OUTCOMES:
Diagnostic accuracy of methods used for VL identification | March 2020 - February 2025
  Evaluation of the diagnostic accuracy of available methods (serological tests, RT-PCR, direct microscopy, and culture) in identifying LV cases, particularly in immunocompromised patients and those with atypical presentations. The study will assess the effectiveness of these tests in different clinical scenarios, including their sensitivity and specificity.
  Measure: Sensitivity, specificity, positive and negative predictive values of diagnostic tests (EIA, IFAT, RT-PCR, rK39 ICT, direct microscopy).
  Unit of measure: Percentage (%). Collection method: Comparison with the diagnostic gold standard (bone marrow biopsy with parasite identification).
Monitoring of therapy tolerability | March 2020 - February 2025
  Ongoing assessment of the safety and tolerability of therapeutic interventions used to treat LV, with a focus on identifying potential adverse effects or complications arising from current treatment regimens. This includes monitoring for any therapy-related side effects and evaluating the suitability of treatment options in different patient populations.
  Measure: Number of participants with adverse events (evaluated according to CTCAE v4.0 criteria).
  Unit of measure: Number of adverse events (n), percentage (%). Collection method: Adverse event reporting forms and clinical reports.
Evaluation of therapeutic outcomes of treated cases. | March 2020 - February 2025
  Comprehensive assessment of the therapeutic outcomes in patients treated for LV, measuring the effectiveness of current treatment protocols in terms of clinical improvement, survival rates, and relapse prevention. This will also involve tracking long-term patient recovery and any subsequent need for retreatment.
  Measure: Complete cure rate, recurrence rate at 6 and 12 months, disease-related mortality.
  Unit of measure: Percentage (%), time to recurrence in days (d). Collection method: Clinical and laboratory follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Viale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - Ospedale M. Bufalini di Cesena, AUSL della Romagna, Cesena, Forlì-Cesena
  - Ospedale G.B. Morgagni L. Pierantoni di Forlì, Forlì, Forlì-Cesena
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Ospedale S. Maria delle Croci di Ravenna, AUSL della Romagna, Ravenna
  - Ospedale Infermi di Rimini, AUSL della Romagna, Rimini

IPD SHARING:
Plan to Share IPD: No